CLINICAL TRIAL: NCT00223327
Title: Measurement of Bite Force in Humans
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 023-1904-101
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Dental Pulp Necrosis; Periapical Periodontitis
Keywords: pain; Normal pulp and normal periodontal status; Chronic apical periodontitis of pulpal origin
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is for a clinical trial to evaluate the reliability of the bite fork as a diagnostic instrument in subjects with pulpal necrosis and apical periodontitis.

DETAILED DESCRIPTION:
This clinical trial consists of two parts. We will first use the bite fork in normal volunteers to evaluate its test-retest and inter-rater reliability. We will then use the bite fork in subjects with differing endodontic diagnoses and compare these results with the standard clinical diagnostic test (percussion).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 16 years of age.
2. Clinical indication for non-surgical root canal therapy (NSRCT).
3. 1st or 2nd maxillary or mandibular molar or premolar
4. Diagnosis must be chronic apical periodontitis (CAP) with or without symptoms.
5. Intact, mature apices.
6. American Society of Anesthesiologists (ASA) I or II.

Exclusion Criteria:

1. Failure to meet any of the above
2. Previous NSRCT
3. Previous pulpotomy or pulpectomy
4. Suppurative apical periodontitis
5. Patients taking medications which can affect their pain rating or medications which affect their immune system (such as glucocorticoids)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Normal subjects and patients with orofacial pain presenting in the dental clinic.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asma A Khan, Principal Investigator — University of Texas Health Science Center at San Antonio, Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States